CLINICAL TRIAL: NCT04082780
Title: A Double-Blind Randomized Placebo-Controlled Trial of Rifamycin SV MXX in Minimal Hepatic Encephalopathy (RIVET Trial)
Brief Title: Rifamycin in Minimal Hepatic Encephalopathy
Acronym: RIVET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAJAJ0025
Record Dates: First submitted 2019-08-22; First posted 2019-09-09 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Hepatic Encephalopathy; Cirrhosis, Liver
Keywords: brain MRI; cognitive testing; microbiota; metabolomics; pharmacokinetics
MeSH Terms: conditions — Hepatic Encephalopathy; Liver Cirrhosis | interventions — rifamycin SV

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomized 1:1 into receiving rifamycin or placebo by a random number generator created by Cosmo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rifamycin (Experimental): Rifamycin-SV MMX 600 mg PO two times a day (1200 mg) for 30 days
  Interventions: Drug: Rifamycin SV MMX
- Placebo (Placebo Comparator): Placebo PO two times a day for 30 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rifamycin SV MMX — Intervention arm
  Other Names: Aemcolo
  Arms: Rifamycin
Other: Placebo — Placebo arm
  Arms: Placebo

SUMMARY:
This is a randomized double-blind placebo-controlled trial of MHE in patients with cirrhosis using rifamycin SV-MMX 600mg BID vs placebo for 30 days with PK, safety, microbiota, brain function and brain MRI endpoints.

DETAILED DESCRIPTION:
Hepatic encephalopathy (HE) is a highly prevalent neuro-cognitive complication of cirrhosis characterized by cognitive dysfunction, and high rate of subsequent mortality and recurrence. HE also places a tremendous burden with a relentless increase in inpatient stay duration with charges topping $7244.7 million in 20092. There were almost 23,000 hospitalizations for HE in 2009 and far more patients with HE who are being managed as an outpatient in the US. In the NACSELD (North American Consortium for the Study of End-Stage Liver Disease) experience, HE in inpatients is an independent risk factor for mortality and the leading cause of readmissions in patients with cirrhosis.

HE has two major phases, covert or minimal HE (MHE), which is only recognized by specialized tests and overt HE (OHE), which is clinically obvious. OHE forms the tip of the iceberg, while MHE affects as many as 60% of tested patients with cirrhosis.

MHE is associated with changes in specific cognitive domains that result in altered health-related quality of life and daily function. This can promote the development of OHE, impair driving and employment, increase falls and is independently associated with a risk of hospitalizations and mortality.

There is an alteration of gut microbial composition and function (bile acid changes, endotoxemia and gut metabolic products) in cirrhosis, which worsens with disease progression with MHE and OHE. Current treatments for OHE are mostly focused on the gut, including lactulose and rifaximin. However, despite extracting a major toll on disease progression, there is no current guideline to treat MHE. Prior studies using lactulose and rifaximin have been performed in this setting with improvement in brain function, brain MRI changes and microbial function. However, these are still not standard of care.

Rifamycin SV MMX® 200 mg is a gut-specific antibiotic with a long track record of safety that has been FDA approved for the treatment of traveler's diarrhea. Unlike rifaximin, rifamycin-SV MMX mostly affects the colon, where the bacterial load is much larger than in the other parts of the GI tract. The impact of rifamycin on MHE has not been studied to date. This is a randomized double-blind placebo-controlled trial of MHE in patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. Cirrhosis defined by any one of the following

   1. Cirrhosis on liver biopsy or transient elastography
   2. Nodular liver on imaging
   3. Endoscopic or radiological evidence of varices in a patient with chronic liver disease
   4. Platelet count <150,000/mm3 and AST/ALT ratio >1 in a patient with chronic liver disease
3. Women of childbearing age will need to be on accepted birth control for 10 days prior to entering study and 30 days after the end of the last dose of the study drug.
4. Cognitive impairment on PHES aggregate score [more than or greater than] -4SD or EncephalApp Stroop - based on norms published in Allampati et al located at the website www.encephalapp.com17 (This is the accepted diagnosis of minimal HE.)
5. Willing and able to participate, provide samples and complete follow-up
6. Stable Liver function tests between 2-12 weeks prior to enrollment (can include the screening laboratory values details in exclusion criteria)

Exclusion Criteria:

1. Unclear diagnosis of cirrhosis (does not meet the criteria outlined above)
2. Child score >8
3. Increasing trend of ALT and AST in the 2-12 weeks prior to study inclusion (Baseline values established by at least two samples obtained at least 2 weeks and no more than 8-12 weeks apart) to account for disease related changes in liver enzymes and bilirubin while on study that may otherwise be inappropriately attributed to study drug. >20% increase in baseline serum AST, ALT, ALP and total bilirubin (TBL) will be considered an exclusion criterion.
4. Unable to consent, follow for the study duration
5. Normal performance on PHES
6. Mini-mental status exam<2518
7. Recent alcohol abuse (within 3 months)
8. Recent illicit drug abuse (within 3 months) except marijuana
9. Current use of psychoactive drugs apart from long-standing opioids or stable anti-depressant use.
10. Prior overt HE episodes defined as West-Haven Criteria grade 2 or higher in the past that required hospitalization or initiation of lactulose or rifaximin therapy
11. Currently on lactulose or rifaximin
12. Current or recent invasive bacterial or fungal infections (<1 month)
13. Allergic reactions to rifamycin, rifampin or rifaximin
14. MELD >20
15. TIPS placement
16. Serum sodium<125
17. On SBP prophylaxis
18. Post-transplant cirrhosis
19. Infections within 4 weeks
20. End-stage organ failures: CHF with EF<25%, End-stage renal disease on dialysis, COPD on home oxygen
21. Pregnancy (positive urine pregnancy test at screening)
22. In the opinion of the PI, those who are unlikely to survive or remain without liver transplant for 6 weeks, or cannot adhere to the trial activities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Cirrhosis Dysbiosis Ratio of stool microbiota | 30 days
  Comparing this ratio in rifamycin compared to placebo groups (Lachnospiraceae + Ruminococcaceae + Clostridium Cluster XIV + Veillonellaceae / Enterobacteriaceae + Bacteroidaceae)

SECONDARY OUTCOMES:
Psychometric hepatic encephalopathy score (PHES) composite score ranges from -15 to +5 | 30 days
  Battery of 5 cognitive tests that yield a numeric composite score. Investigators will compare this score in rifamycin compared to placebo groups. Higher total score = better performance. Norms are at www.encephalapp.com, which are adjusted for age, gender and education status.
EncephalApp Stroop OffTime+OnTime is the total time taken to complete 5 runs in Off and 5 runs in On state. | 30 days
  Cognitive test. Investigators will compare this score in rifamycin compared to placebo groups. High score = worse performance. Norms are at www.encephalapp.com, which are adjusted for age, gender and education status.
Sickness Impact Profile total score is the total score determined after all 12 domains are scored | 30 days
  Validated questionnaire for health-related quality of life. Investigators will compare this score in rifamycin compared to placebo groups. There is no defined range but a higher score indicates worse QOL.
Sickness Impact Profile psychosocial score is the score of the psychosocial part of the SIP | 30 days
  Validated questionnaire for health-related quality of life. Investigators will compare this score in rifamycin compared to placebo groups. There is no defined range but a higher score indicates worse QOL.
Sickness Impact Profile physical score is the score of the physical part of the SIP | 30 days
  Validated questionnaire for health-related quality of life. Investigators will compare this score in rifamycin compared to placebo groups.There is no defined range but a higher score indicates worse QOL.
Pittsburgh sleep quality index | 30 days
  Validated questionnaire for sleep quality. Investigators will compare this in rifamycin compared to placebo groups
Serious adverse events (Hospitalizations, death, prolongation of hospitalizations) | 30 days
  Investigators will compare this in rifamycin compared to placebo groups
Serious adverse events (Hospitalizations, death, prolongation of hospitalizations) | 37 days
  Investigators will compare this in rifamycin compared to placebo groups
Adverse events related to rifamycin | 30 days
  Investigators will compare this in rifamycin compared to placebo groups
Adverse events related to rifamycin | 37 days
  Investigators will compare this in rifamycin compared to placebo groups
Systemic exposure of rifamycin in the blood | Baseline
  AUC of rifamycin levels in the 6 hourly blood collection time-points post rifamycin ingestion will be studied on day 1
Systemic exposure of rifamycin in the blood | 15 days
  Spot plasma level of rifamycin will be analyzed
Systemic exposure of rifamycin in the urine | Baseline
  AUC of rifamycin levels in the 6 hours urine collection post rifamycin ingestion will be studied on day 1
Systemic exposure of rifamycin in the urine | 15 days
  Spot urine level of rifamycin will be analyzed
Untargeted Metabolomics in serum using LC/MS | 30 days
  Investigators will compare these in rifamycin compared to placebo groups
Calprotectin levels in stool | 30 days
  Investigators will compare these in rifamycin compared to placebo groups
Untargeted Metabolomics in urine using LC/MS | 30 days
  Investigators will compare these in rifamycin compared to placebo groups
Fecal bile acid levels | 30 days
  Using LC/MS. Investigators will compare these in rifamycin compared to placebo groups
Microbiota diversity using Shannon index | 30 days
  Stool microbiota diversity. Investigators will compare these in rifamycin compared to placebo groups ranges widely from 0-20

OTHER OUTCOMES:
Handgrip strength | 30 days
  Jamar hand dynanometer; Investigators will compare these in rifamycin compared to placebo groups
Body Muscle composition | 30 days
  InBody assessment; Investigators will compare these in rifamycin compared to placebo groups
Brain MR Spectroscopy in Anterior cingulate cortex, posterior gray matter, and right parietal white matter in a subset | 30 days
  Investigators will compare these in rifamycin compared to placebo groups and measure choline, GSH, glutamate/glutamine and myoinositol

CONTACTS AND LOCATIONS:
Overall Officials: JASMOHAN BAJAJ, Principal Investigator — Hunter Holmes McGuire Medical Center
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No